CLINICAL TRIAL: NCT03781349
Title: Comparative Efficacy on Pain of Two Non-pharmacological Treatments (TENS or MENS) in Patients With Partial Rotator Cuff Tears. A Randomized Trial
Brief Title: TENS of MENS for Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Assistant Professor of Anesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBD624/6-2-15
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MENS (Active Comparator): MENS are applied through placement of six electrodes (size of 4x4cm), of which four were placed exactly like the TENS electrodes and the other two, one in the palm and the other at the height of the asteroid ganglion. Duration of the intervention was 24 min for a total of 15 sessions. The frequency was 50 Hz and the intensity was 100 μA.
  Interventions: Device: MENS
- TENS (Active Comparator): TENS are applied through the placement of four electrodes on either side of the deltoid muscle, on the front and back surfaces of the shoulder joint for 20 min and each patient received 15 sessions (five per week). A constant current of high frequency was used (100 HZ) and its intensity was initiated at 10mA and was then gradually increased to 15mA
  Interventions: Device: TENS

INTERVENTIONS:
Device: MENS
  Arms: MENS
Device: TENS
  Arms: TENS

SUMMARY:
The aim of this study was to clarify the effectiveness of physiotherapeutic intervention through the TENS or MENS in conjunction with kinesiotherapy in patients with partial thickness rotator cuff tear.

DETAILED DESCRIPTION:
The primary characteristic of a rotator cuff tear is pain, while muscle weakness appears as a secondary feature, leading to further disability.

The aim of this study was to clarify the effectiveness of physiotherapeutic intervention through the TENS or MENS in conjunction with kinesiotherapy in patients with partial thickness rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering shoulder pain because of partial thickness rotator cuff tear, confirmed with MRI and ultrasound scanning.
* Patients not receiving any recent pharmacotherapy with NSAIDs during the last month, or surgery at the shoulder area at any time point,
* The referral orthopedic had suggested physiotherapy.

Exclusion Criteria:

* Patients with open wounds or skin diseases in the shoulder area
* pregnant women
* patients with any type of neoplastic disease
* patients with pacemakers or serious cardiovascular diseases including arrhythmia, - patients with collagen diseases
* history of shoulder surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity: NRS | up to 3 months after intervention
  Numeric Rating Scale, ranging from 0-10 (with 0 = no pain, and 10=worst pain). It measures pain intensity
Disability | up to 3 months after intervention
  SPADI questionnaire (shoulder pain and disability questionnaire). It measures pain and disability caused by shoulder diseases, each question ranging between 0 and 10 (with 0 indicating no disability and 10 indicating worst disability). It includes 5 questions about pain and 8 questions about disability.

SECONDARY OUTCOMES:
quality of patients' life: EQ 5D | up to 3 months after intervention
  EQ 5D, EuroQol measuring of perceived Health today, Scale 0-100 (with 0 indicating worst health, and 100 indicating best imaginable health as perceived by the patient)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided